CLINICAL TRIAL: NCT00921193
Title: Evaluation of Radiation Therapy Positioning System (RTPS) in Patients With Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navotek Medical, Ltd. (Industry)
Responsible Party: Tal Shchory, COO, Navotek Medical ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-14-001
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer
Keywords: Prostate; fiducials; radiation Therapy; Tracking; Localization
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Radiation Therapy Positioning System (RTPS)

SUMMARY:
The study aims to evaluate the safety and performance of the RTPS in patients with localized prostate cancer.The RTPS is an investigational device and requires permanent implantation of a small radioactive fiducial, called the Blip, in the prostate.

DETAILED DESCRIPTION:
The high precision of planned radiotherapy treatments requires accurate positioning of the prostate in order to ensure that the tightly conformed dose distribution does not miss the prostate and result in either significant tumor underdosage, an increased dose to the rectum or bladder, or both. Precise delivery has been addressed using a variety of pre-treatment localization systems. The most direct localization of the prostate involves the use of ultrasound, computed tomography (CT), or radiography of permanently implanted fiducial markers.

In this study the safety and performance of a novel investigational tracking system will be evaluated. The Radiation Therapy Positioning System (RTPS) is a radioactive tracking system integrated into the radiotherapy set-up workflow. The System is composed of the Clinical Positioning System (CPS) and a radioactive soft tissue implanted fiducial (Blip), which is permanently implanted in the prostate. By tracking the implanted Blip, the CPS can monitor positional changes prior to and during the treatment.

The accuracy of the RTPS localization will be compared to the CBCT in at least 5 radiation therapy sessions per patient.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of adenocarcinoma of the prostate.
2. Male, age greater than or equal to 45 years.
3. Intact prostate of at least 30g, as estimated by physical estimation and/or ultrasound.
4. ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
5. Patients must be planned to have external beam radiation as the definitive treatment for their prostate cancer with treatment set-up verification according to a locally fixed protocol.
6. Patients must have anatomy that will allow an adequate pelvic imaging by CBCT as well as CT scanning.
7. Organ confined or locally advanced prostate cancer with clinical N category 0 or x, M category 0 or x.
8. Ability to comply with study visit schedule.
9. Patient (or legal guardian) understands the study requirements and the investigational procedure and provides written Informed Consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

1. Past history of abdominoperineal (A-P) resection.
2. Planned course of treatment using brachytherapy (permanent brachytherapy seeds or high dose rate [HDR] brachytherapy).
3. Allergy to local anesthetics.
4. History of chronic prostatitis.
5. Patients with history of recent acute and/or chronic bleeding disorders.
6. Patients on therapeutic anti-coagulants or anti-platelet therapy, not including aspirin or dipyridamole.
7. Patients for which the maximum body width or the maximum anterior-posterior depth in the abdomino-pelvic region is greater than 40 cm. (Measurements will be made visually with a ruler.)
8. Patients with a body habitus that the CT bore of the CT/LINAC treatment machine cannot accommodate.
9. Patients with a prior history of pelvic or prostate radiotherapy.
10. Patients who have had prior prostate surgery other than a TUR.
11. Cognitively impaired patients who cannot give informed consent.
12. Patients with hip replacement by a metal prosthesis.
13. Patient has participated in, or is planned to participate in, any investigational drug or device study within the past or next 2 months.
14. Patient who has more than 1μCi of any injected or implanted radioactive material within his body.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Device related adverse events by evaluation of the type, frequency and severity of the device, implantation device and/or implantation procedure related adverse events | 6 months
International Prostate Symptom Score (IPSS) questionnaire at baseline, at CT planning and on first week of Radiation Therapy. | 3 weeks
Successful implantation of the Blip in the prostate | 1 wk
Non migration of the Blip as evaluated by measuring the average absolute change in inter-marker distances measured during and at the end of radiotherapy treatment | 10 weeks
Performance of the RTPS in at least five of approximately 40 radiation therapy sessions | 8 weeks

SECONDARY OUTCOMES:
Record target volume movement during at least 5 radiation therapy sessions | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip MP Poortmans, MD, PhD, Principal Investigator — Dr. Bernard Verbeeten Instituut; Willy JM de Kruijf, PhD, Principal Investigator — Dr. Bernard Verbeeten Instituut; Karin Haustermans, MD, Principal Investigator — Leuvens Kankerinstituut
Locations (2):
- Leuvens Kankerinstituut, Leuven, Belgium
- Dr. Bernard Verbeeten Institute, Tilburg, Netherlands

REFERENCES:
- See also: sponsor's website — http://www.navotek.com